CLINICAL TRIAL: NCT02483416
Title: Evaluation of the Impact of a Nurse-led Telephone Follow-up on Treatment Compliance of Patients Treated From a Locally Advanced or Metastatic Non-small-cell Lung Cancer (NSCLC) With Activating Epidermal Growth Factor Receptor (EGFR) Mutation(s).The PARTAGE Study.
Brief Title: Evaluation of the Impact of Nurse-led Telephone on Treatment Compliance
Status: Terminated | Type: Observational
Why Stopped: Poor recruitment
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200.227
Record Dates: First submitted 2015-04-09; First posted 2015-06-26 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2018-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- group 1: Group without 'remote additional personalised nurse-led follow-up: patients will receive the healthcare given routinely by their medical team
- group 2: Group with 'remote additional personalised nurse-led follow-up: patients will receive telephone calls from a nurse in addition to the healthcare given routinely by their medical team

SUMMARY:
The study will take place over a period of 27 months. The recruitment phase will last approximately 24 months and each patient will participate for approximately 3 months.

At the inclusion visit (D0), the investigator will ask the patient whether he would like to participate in the study and will obtain his written consent.

Patients agreeing to participate will be randomised (3:1 ratio) and included in one of the following 2 groups:

Group without 'remote additional personalised nurse-led follow-up: patients will receive the healthcare given routinely by their medical team (100 patients).

Group with 'remote additional personalised nurse-led follow-up: patients will receive telephone calls from a nurse in addition to the healthcare given routinely by their medical team (300 patients).

All the patients will be seen according to normal practice by the study medical team.

Patients in the group with 'remote additional personalised nurse-led follow-up will be contacted 8 times during the study (at D1, D7, D14, D21, D28, D44, D59 and D89). The nurse will make sure that the treatment takes place in good conditions; she cannot intervene in the medical care of the patient, nor give answer to the questions relative to the disease or to the treatment of the patient. The medical team remains the privileged contact of the patient.

DETAILED DESCRIPTION:
Purpose:

Study Design:

ELIGIBILITY:
Inclusion criteria:

Male or female patient older than 18 years. Adult patient diagnosed with stage IIIb/IV NSCLC locally advanced or metastatic, with activating mutation(s) of EGFR and who is EGFR-TKI naïve.

Patient for whom a decision of treatment with afatinib monotherapy has been taken in the frame of its marketing authorization.

Out-patient. Patient having given written consent for participation in the study. Patient who is able to participate in the investigator's opinion. Patient affiliated with the French social security.

Exclusion criteria:

Patients participating in an interventional clinical study. Patients for whom a participation in an interventional clinical study is foreseen within 3 months following the study inclusion.

Patients participating in a therapeutic education program.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC EGFR mutated
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (34):
- France (34):
  - CLI Dr Calabet, Oncolgie, Agen, Agen
  - HOP Centre Hospitalier Pays d'Aix, Pneumo, Aix en Provence, Aix-en-Provence
  - CLI Polyclinique du Parc Rambot, Pneumo, Aix en Provence, Aix-en-Provence
  - HOP Centre Marie Curie, Onco, Arras, Arras
  - HOP Centre Hospitalier de Béziers, Pneumo, Béziers, Béziers
  - CLI Bordeaux Nord Aquitaine, Bordeaux
  - CLI Tivoli, Bordeaux
  - CH, Oncologie, Brive la Gaillarde,, Brive-la-Gaillarde
  - HOP Louis Pradel, Bron
  - CLI du Parc, Pneumo, Castelnau le Lez, Castelnau-le-Lez
  - Centre médical N de Pontoux, Oncologie, Chalon sur Saône, Chalon-sur-Saône
  - HOP de Chauny, Chauny
  - Centre Hospitalier Intercommunal, Oncolgie, Crétail, Créteil
  - HOP La Dracénie, Onco, Draguignan, Draguignan
  - HOP CHD La Roche sur Yon - Montaigu - Luçon, Pneumo, La Roche-sur-Yon
  - HOP CH Emile Roux Le Puy, Pneumo, Le puy en Velay, Le Puy-en-Velay
  - HOP Hôpital Robert Boulin, Pneumo, Libourne, Libourne
  - Hopital Privé Jean Mermoz, Lyon
  - HOP Saint Joseph et Saint Luc, Pneumo, Lyon, Lyon
  - CHG, Oncologie, Meaux, Meaux
  - CLI Clémentville, Montpellier
  - HOP Centre Hospitalier de Mulhouse, Pneumo, Mulhouse, Mulhouse
  - CTR d'Oncologie de Gentilly, Onco, Nancy, Nancy
  - CLI Polyclinique le Languedoc, Narbonne, Narbonne
  - CLI Saint-Pierre, Oncologie, Perpignan, Perpignan
  - CHR d'Annecy, Oncologie, Annecy, Pringy
  - HOP Cornouaille, Pneumo, Quimper, Quimper
  - CLI Les Bleuets, Pneumologie, Reims, Reims
  - HOP Centre Hospitalier de Saint Quentin, Pneumo, St-Quentin, Saint-Quentin
  - HOP Hôpitaux du Léman, Thonon-les-Bains
  - HOP HIA Saint-Anne, Toulon
  - CLI Pasteur, Toulouse
  - Centre de Radiothérapie Marie Curie, Valence
  - HOP Nord Ouest de Villefranche, oncologie, Gleize, Villefranche-sur-Saône

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 14 French active centres and lasted 14 months. The recruitment phase was stopped after 10.7 months. Each patient participated for approximately 3 months. Actual subjects enrolled were 30 but two subjects are not included because of incomplete case record form (CRF)
Pre-assignment Details: Patients for whom a decision of treatment with afatinib monotherapy has been taken in the frame of its marketing authorization were included in this trial.
Groups:
- Group With Nurse-led Telephone Follow-up: Group with remote additional personalised nurse-led follow-up: patients received telephone calls from a nurse in addition to the healthcare given routinely by their medical team
- Group Without Nurse-led Telephone Follow-up: Group without remote additional personalised nurse-led follow-up: patients received the healthcare given routinely by their medical team
Period: Overall Study
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Started | 21 | 7
Completed | 18 | 6
Not Completed | 3 | 1
Not completed — Other reason | 0 | 1
Not completed — Treatment stop | 3 | 0

BASELINE CHARACTERISTICS:
Population: Randomised patients who satisfy the essential inclusion and exclusion criteria, and for whom information is available for the major evaluation criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up | Total
Number analyzed (Participants) | 21 | 7 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (10.9) | 69.9 (12.6) | 65.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 3 | 19
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Cumulated Dose Milligram (mg) of Oral Targeted Therapy During the 3-month Follow-up.
Description: The cumulated dose (mg) of oral targeted therapy taken between visits is the sum of the doses (mg) of the tablets taken by the patient. The cumulated dose (mg) of the oral targeted therapy taken during the 3-month follow-up is the sum of the doses (mg) cumulated taken between visits during the 3-month follow-up.
Time Frame: 3 months
Population: The primary analysis population will be the population of randomised patients who satisfy the essential inclusion and exclusion criteria, and for whom information is available for the major evaluation criteria (in particular the primary criterion)- Observed cases
Measure: Median (Full Range); unit: milligram (mg)
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 5 | 2
milligram (mg) | 3120 [2350 to 3680] | 3220.0 [3080 to 3360]

2. Secondary Outcome: Score (0-6) Obtained With the Girerd Questionnaire
Description: Girerd questionnaire is a questionnaire composed of 6 binary questions (yes/no) and is used to assess treatment compliance. The final score obtained is the number of questions to which the patient responded "yes". Thus, the score ranges from 0 to 6. A patient will be classified as:
  Good compliant with score = 0. Minor non-compliant with score = 1 or 2. Non-compliant with score >2.
Time Frame: at Day 30 (D30), Day 60 (D60) and Day 90 (D90)
Population: Population of randomised patients who satisfy the essential inclusion and exclusion criteria, and for whom information is available for the major evaluation criteria (in particular the primary criterion)- Observed cases
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7
scores on a scale
  D30: number analyzed (Participants) | 16 | 6
  D30 | 0.3 (0.6) | 0.0 (0.0)
  D60: number analyzed (Participants) | 16 | 3
  D60 | 0.4 (0.6) | 0.0 (0.0)
  D90: number analyzed (Participants) | 15 | 5
  D90 | 0.4 (0.6) | 0.2 (0.4)

3. Secondary Outcome: Cumulated Dose of Oral Targeted Therapy Not Taken (All Categories) Following Decision of the Medical Team
Description: The cumulated dose (mg) of oral targeted therapy not taken between 2 visits is the sum of the doses (mg) of tablets not taken by the patient. The cumulated dose (mg) of oral targeted therapy not taken during the 3-month follow-up is the sum of the cumulated doses (mg) not taken between 2 visits during the 3-month follow-up.
Time Frame: 3 months
Population: as for outcome 1
Measure: Median (Full Range); unit: milligram (mg)
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 4 | 2
milligram (mg) | 520 [0 to 800] | 420 [80 to 760]

4. Secondary Outcome: Cumulated Dose of Oral Targeted Therapy Not Taken Due to Dose Reduction Following Decision of the Medical Team.
Description: Cumulated dose of oral targeted therapy not taken due to dose reduction following decision of the medical team.
  There were no participants with dose reduction hence the data is not available.
Time Frame: 3 months
Population: as for outcome 1
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Cumulated Dose of Oral Targeted Therapy Not Taken Due to Temporary or Definitive Interruption Following the Medical Team Decision.
Description: Cumulated dose of oral targeted therapy not taken due to temporary or definitive interruption following the medical team decision.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram (mg)
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7
milligram (mg)
  Temporary interruption: number analyzed (Participants) | 1 | 0
  Temporary interruption | 0.0 (NA) — As only 1 participant hence the standard deviation is not available |
  Definitive interruption: number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Cumulated Dose of Oral Targeted Therapy Not Taken (All Categories) Following Patient Decision.
Description: Cumulated dose of oral targeted therapy not taken (all categories) following patient decision. Cumulated dose not taken in total is missing since no patient without therapy following patient decision
Time Frame: 3 months
Population: as for outcome 1
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Cumulated Dose of Oral Targeted Therapy Not Taken Due to Dose Reduction Following Patient Decision.
Description: Cumulated dose of oral targeted therapy not taken due to dose reduction following patient decision. No participants with dose reduction.
Time Frame: 3 months
Population: The primary analysis population will be the population of randomised patients who satisfy the essential inclusion and exclusion criteria, and for whom information is available for the major evaluation criteria (in particular the primary criterion)- only participants with dose reduction
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Cumulated Dose of Oral Targeted Therapy Not Taken Due to Temporary or Definitive Interruption Following Patient Decision.
Description: Cumulated dose of oral targeted therapy not taken due to temporary or definitive interruption following patient decision.
  No patient without therapy following patient decision
Time Frame: 3 months
Population: The primary analysis population will be the population of randomised patients who satisfy the essential inclusion and exclusion criteria, and for whom information is available for the major evaluation criteria (in particular the primary criterion)
Measure: Mean (Standard Deviation); unit: milligram (mg)
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7

9. Secondary Outcome: Visual Analogue Scale (VAS) Score (0-10) for Overall Patient Satisfaction With the Level of Care (Information, Advice) at D90.
Description: VAS scores will be presented in the form of a horizontal ungraduated line of 10 centimeters (cm), with the following extremities: left, 'completely unsatisfied' and right, 'very satisfied'. The number of points (0 to 10) obtained in VAS corresponds to the distance (cm) between the left extremity of the line and the mark placed on the line by the patient, investigator, general practitioner, or pharmacist to assess patient's level of satisfaction.
Time Frame: 3 months
Population: as for outcome 8
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 15 | 5
scores on a scale | 9 [2 to 10] | 10 [5 to 10]

10. Secondary Outcome: Change in Quality of Life Questionnaire Functional Assessment of Cancer Therapy Lung (FACT-L) Score Between D30 and D0, Between D90 and D30 and Between D90 and D0
Description: The patients' quality of life was evaluated with the FACT-L questionnaire. This questionnaire explores 4 dimensions of well-being: physical, social and emotional. These items are completed by 9 questions specific to lung cancer. Subscale scores are added to obtain total score. Scores obtained with this questionnaire range between 0 and 136. The higher the score the better the quality of life.
Time Frame: Day0 (D0), Day30 (D30) and Day90 (D90)
Population: as for outcome 8
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7
scores on a scale
  Absolute variation between D30 and D0: number analyzed (Participants) | 15 | 5
  Absolute variation between D30 and D0 | -4 [-41 to 14] | 1 [-8 to 60]
  Absolute variation between D90 and D0: number analyzed (Participants) | 12 | 5
  Absolute variation between D90 and D0 | -8 [-31 to 18] | 4 [-3 to 54]
  Absolute variation between D90 and D30: number analyzed (Participants) | 12 | 4
  Absolute variation between D90 and D30 | -2 [-31 to 27] | 0 [-7 to 6]

11. Secondary Outcome: Number of Emergency Admissions (Related to the Treatment) During the 3-month Follow-up.
Description: Number of participants with emergency admissions (related to the treatment) during the 3-month follow-up are presented
Time Frame: Day30 (D30), Day60 (D60) and Day90 (D90)
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7
Participants
  D30- no admission: number analyzed (Participants) | 19 | 6
  D30- no admission | 18 | 5
  D30- 1 admission: number analyzed (Participants) | 19 | 6
  D30- 1 admission | 1 | 1
  D60- no admission: number analyzed (Participants) | 17 | 5
  D60- no admission | 14 | 5
  D60- 1 admission: number analyzed (Participants) | 17 | 5
  D60- 1 admission | 3 | 0
  D90- no admission: number analyzed (Participants) | 18 | 5
  D90- no admission | 17 | 4
  D90- 1 admission: number analyzed (Participants) | 18 | 5
  D90- 1 admission | 1 | 1

12. Secondary Outcome: Number of Unplanned Hospitalizations (Related to the Treatment) During the 3-month Follow-up
Description: Number of participants with unplanned hospitalizations (related to the treatment) during the 3-month follow-up is presented
Time Frame: D30, D60, D90
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7
Participants
  D30- no hospitalization: number analyzed (Participants) | 19 | 6
  D30- no hospitalization | 18 | 6
  D30- 1 hospitalization: number analyzed (Participants) | 19 | 6
  D30- 1 hospitalization | 1 | 0
  D60- no hospitalization: number analyzed (Participants) | 18 | 5
  D60- no hospitalization | 16 | 5
  D60- 1 hospitalization: number analyzed (Participants) | 18 | 5
  D60- 1 hospitalization | 2 | 0
  D90- no hospitalization: number analyzed (Participants) | 18 | 5
  D90- no hospitalization | 16 | 5
  D90- 1 hospitalization: number analyzed (Participants) | 18 | 5
  D90- 1 hospitalization | 2 | 0

13. Secondary Outcome: Duration of Unplanned Hospitalizations (Related to the Treatment)) During the 3-month Follow-up.
Description: Duration of unplanned hospitalizations (related to the treatment) during the 3-month follow-up are presented
Time Frame: D30, D60 and D90
Population: as for outcome 8
Measure: Median (Full Range); unit: days
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7
days
  D30: number analyzed (Participants) | 1 | 0
  D30 | 13 [13 to 13] |
  D60: number analyzed (Participants) | 1 | 0
  D60 | 3 [3 to 3] |
  D90: number analyzed (Participants) | 2 | 0
  D90 | 14 [4 to 23] |

14. Secondary Outcome: Number of Unplanned Visits to the Investigator During the 3-month Follow-up
Description: Number of participants with unplanned visits to the investigator during the 3-month follow-up are presented
Time Frame: D30, D60 and D90
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7
Participants
  D30- no visit: number analyzed (Participants) | 19 | 6
  D30- no visit | 16 | 6
  D30- 1 visit: number analyzed (Participants) | 19 | 6
  D30- 1 visit | 3 | 0
  D60- no visit: number analyzed (Participants) | 18 | 5
  D60- no visit | 14 | 5
  D60- 1 visit: number analyzed (Participants) | 18 | 5
  D60- 1 visit | 4 | 0
  D90- no visit: number analyzed (Participants) | 18 | 5
  D90- no visit | 17 | 5
  D90- 1 visit: number analyzed (Participants) | 18 | 5
  D90- 1 visit | 1 | 0

15. Secondary Outcome: Number of Unplanned Visits to a Specialist, Whatever is His Specialty, Other Than the Investigator During the 3-month Follow-up.
Description: Number of participants with unplanned visits to a specialist, whatever is his specialty, other than the investigator during the 3-month follow-up is presented
Time Frame: D30, D60 and D90
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7
Participants
  D30- no visit: number analyzed (Participants) | 17 | 6
  D30- no visit | 14 | 6
  D30- 1 visit: number analyzed (Participants) | 17 | 6
  D30- 1 visit | 2 | 0
  D30- 3 visits: number analyzed (Participants) | 17 | 6
  D30- 3 visits | 1 | 0
  D60- no visit: number analyzed (Participants) | 17 | 4
  D60- no visit | 16 | 3
  D60- 1 visit: number analyzed (Participants) | 17 | 4
  D60- 1 visit | 1 | 1
  D90- no visit: number analyzed (Participants) | 17 | 5
  D90- no visit | 15 | 5
  D90- 1 visit: number analyzed (Participants) | 17 | 5
  D90- 1 visit | 1 | 0
  D90- 2 visit: number analyzed (Participants) | 17 | 5
  D90- 2 visit | 1 | 0

16. Secondary Outcome: Number of Unplanned Visits to the General Practitioner During the 3-month Follow-up
Description: Number of participants with unplanned visits to the general practitioner during the 3-month follow-up is presented
Time Frame: D30, D60 and D90
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7
Participants
  D30- no visit: number analyzed (Participants) | 16 | 5
  D30- no visit | 11 | 4
  D30- 1 visit: number analyzed (Participants) | 16 | 5
  D30- 1 visit | 4 | 1
  D30- 2 visits: number analyzed (Participants) | 16 | 5
  D30- 2 visits | 1 | 0
  D60- no visit: number analyzed (Participants) | 16 | 3
  D60- no visit | 13 | 3
  D60- 1 visit: number analyzed (Participants) | 16 | 3
  D60- 1 visit | 3 | 0
  D90- no visit: number analyzed (Participants) | 16 | 5
  D90- no visit | 13 | 3
  D90- 1 visit: number analyzed (Participants) | 16 | 5
  D90- 1 visit | 3 | 2

17. Secondary Outcome: VAS Score (0-10) for Overall Investigator Satisfaction With the Level of Patient Care at D90
Description: VAS score (0-10) for overall investigator satisfaction with the level of patient care at D90 (Overall investigator satisfaction) is presented.
  VAS scores will be presented in the form of a horizontal ungraduated line of 10 centimeters (cm), with the following extremities: left, 'completely unsatisfied' and right, 'very satisfied'. The number of points (0 to 10) obtained in VAS corresponds to the distance (cm) between the left extremity of the line and the mark placed on the line by the patient, investigator, general practitioner, or pharmacist to assess patient's level of satisfaction.
Time Frame: D90
Population: as for outcome 8
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 20 | 6
scores on a scale | 8 [1 to 10] | 7 [6 to 10]

18. Secondary Outcome: VAS Score (0-10) for Overall General Practitioner Satisfaction With the Level of Patient Care at D90 (Only for the Patients With 'Remote Additional Personalised Nurse-led Follow-up)
Description: VAS score (0-10) for overall general practitioner satisfaction with the level of patient care at D90 (only for the patients with 'remote additional personalised nurse-led follow-up) (Overall general practitioner satisfaction) is presented.
  VAS scores will be presented in the form of a horizontal ungraduated line of 10 centimeters (cm), with the following extremities: left, 'completely unsatisfied' and right, 'very satisfied'. The number of points (0 to 10) obtained in VAS corresponds to the distance (cm) between the left extremity of the line and the mark placed on the line by the patient, investigator, general practitioner, or pharmacist to assess patient's level of satisfaction.
Time Frame: D90
Population: as for outcome 8
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 1 | 0
scores on a scale | 8 [8 to 8] |

19. Secondary Outcome: VAS Score (0-10) for Overall Pharmacist Satisfaction With the Level of Patient Care at D90 (Only for the Patients With 'Remote Additional Personalised Nurse-led Follow-up).
Description: VAS score (0-10) for overall pharmacist satisfaction with the level of patient care at D90 (only for the patients with 'remote additional personalised nurse-led follow-up)(Overall pharmacist satisfaction) is presented.
  VAS scores will be presented in the form of a horizontal ungraduated line of 10 centimeters (cm), with the following extremities: left, 'completely unsatisfied' and right, 'very satisfied'. The number of points (0 to 10) obtained in VAS corresponds to the distance (cm) between the left extremity of the line and the mark placed on the line by the patient, investigator, general practitioner, or pharmacist to assess patient's level of satisfaction.
Time Frame: D90
Population: as for outcome 8
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 1 | 0
scores on a scale | 9 [9 to 9] |

20. Secondary Outcome: Number of Calls Made by the Patients to Their General Practitioner During the 3-month Follow-up.
Description: Number of calls made by the patients to their general practitioner during the 3-month follow-up is presented
Time Frame: D30, D60 and D90
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7
Participants
  D30- no call: number analyzed (Participants) | 16 | 5
  D30- no call | 15 | 5
  D30-1 call: number analyzed (Participants) | 16 | 5
  D30-1 call | 1 | 0
  D60- no call: number analyzed (Participants) | 14 | 3
  D60- no call | 12 | 3
  D60-1 call: number analyzed (Participants) | 14 | 3
  D60-1 call | 1 | 0
  D60-3 calls: number analyzed (Participants) | 14 | 3
  D60-3 calls | 1 | 0
  D90- no call: number analyzed (Participants) | 13 | 4
  D90- no call | 13 | 2
  D90-1 call: number analyzed (Participants) | 13 | 4
  D90-1 call | 0 | 2

21. Secondary Outcome: Number of Calls Made by the General Practitioner to the Patient During the 3-month Follow-up.
Description: Number of calls made by the general practitioner to the patient during the 3-month follow-up is presented
Time Frame: D30, D60 and D90
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7
Participants
  D30- no call: number analyzed (Participants) | 15 | 5
  D30- no call | 15 | 5
  D60-no call: number analyzed (Participants) | 15 | 3
  D60-no call | 15 | 3
  D90-no call: number analyzed (Participants) | 14 | 4
  D90-no call | 14 | 4

22. Secondary Outcome: Number of Calls Made by the Patients to Their Medical Team During the 3-month Follow-up
Description: Number of calls made by the patients to their medical team during the 3-month follow-up is presented
Time Frame: D30, D60 and D90
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7
Participants
  D30- no call: number analyzed (Participants) | 19 | 5
  D30- no call | 13 | 4
  D30- 1 call: number analyzed (Participants) | 19 | 5
  D30- 1 call | 4 | 1
  D30- 2 call: number analyzed (Participants) | 19 | 5
  D30- 2 call | 2 | 0
  D60- no call: number analyzed (Participants) | 17 | 4
  D60- no call | 13 | 4
  D60- 1 call: number analyzed (Participants) | 17 | 4
  D60- 1 call | 3 | 0
  D60- 2 call: number analyzed (Participants) | 17 | 4
  D60- 2 call | 1 | 0
  D90- no call: number analyzed (Participants) | 16 | 4
  D90- no call | 15 | 4
  D90- 1 call: number analyzed (Participants) | 16 | 4
  D90- 1 call | 1 | 0

23. Secondary Outcome: Number of Calls Made by the Medical Team to Their Patient During the 3-month Follow-up
Description: Number of calls made by the medical team to their patient during the 3-month follow-up is presented
Time Frame: D30, D60 and D90
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7
Participants
  D30- no call: number analyzed (Participants) | 16 | 5
  D30- no call | 10 | 3
  D30- 1 call: number analyzed (Participants) | 16 | 5
  D30- 1 call | 2 | 2
  D30- 2 calls: number analyzed (Participants) | 16 | 5
  D30- 2 calls | 2 | 0
  D30- 3 calls: number analyzed (Participants) | 16 | 5
  D30- 3 calls | 2 | 0
  D60- no call: number analyzed (Participants) | 17 | 4
  D60- no call | 11 | 4
  D60- 1 call: number analyzed (Participants) | 17 | 4
  D60- 1 call | 3 | 0
  D60- 2 calls: number analyzed (Participants) | 17 | 4
  D60- 2 calls | 1 | 0
  D60- 3 calls: number analyzed (Participants) | 17 | 4
  D60- 3 calls | 2 | 0
  D90- no call: number analyzed (Participants) | 16 | 5
  D90- no call | 14 | 4
  D90- 1 call: number analyzed (Participants) | 16 | 5
  D90- 1 call | 2 | 1

24. Secondary Outcome: Number of Calls Between the General Practitioners and the Medical Teams During the 3-month Follow-up
Description: Number of calls between the general practitioners and the medical teams during the 3-month follow-up is presented
Time Frame: D30, D60, D90
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7
Participants
  D30- no call: number analyzed (Participants) | 13 | 5
  D30- no call | 13 | 5
  D60- no call: number analyzed (Participants) | 11 | 3
  D60- no call | 11 | 3
  D90- no call: number analyzed (Participants) | 15 | 5
  D90- no call | 15 | 4
  D90- 1 call: number analyzed (Participants) | 15 | 5
  D90- 1 call | 0 | 1

25. Secondary Outcome: Number of Adverse Events (AEs), of AEs of Grade ≥ 3, of SAEs Related to the Oral Biological Therapy and Number of AEs Related to the Oral Targeted Therapy Which Causes Temporary or Definitive Discontinuation of the Treatment or Dose Reduction.
Description: Number of participants with Adverse events AEs, of AEs of grade ≥ 3, of serious adverse events (SAEs) related to the oral biological therapy and Number of AEs related to the oral targeted therapy which causes temporary or definitive discontinuation of the treatment or dose reduction are presented
Time Frame: up to 3 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up
Number analyzed (Participants) | 21 | 7
Participants
  Adverse events (AEs) | 21 | 6
  AEs of grade ≥3 | 6 | 1
  SAEs related to oral biological therapy | 2 | 1
  AEs related to oral targeted therapy | 21 | 6

ADVERSE EVENTS:
Time Frame: All Adverse events occurring during the course of the study (i.e., from signing the informed consent onwards through Day 90)
Groups:
- Total: Total of reporting groups
Arm/Group | Group With Nurse-led Telephone Follow-up | Group Without Nurse-led Telephone Follow-up | Total
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/7 | 0/28
Serious Adverse Events (participants affected / at risk) | 2/21 | 1/7 | 3/28
Other Adverse Events (participants affected / at risk) | 21/21 | 6/7 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group With Nurse-led Telephone Follow-up (N=21) | Group Without Nurse-led Telephone Follow-up (N=7) | Total (N=28)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1
Transaminases increased (Investigations) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group With Nurse-led Telephone Follow-up (N=21) | Group Without Nurse-led Telephone Follow-up (N=7) | Total (N=28)
Diarrhoea (Gastrointestinal disorders) | 17 | 4 | 21
Nausea (Gastrointestinal disorders) | 4 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2
Faces soft (Gastrointestinal disorders) | 2 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 2
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 3 | 11
Rash (Skin and subcutaneous tissue disorders) | 8 | 3 | 11
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 | 0 | 5
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Fatigue (General disorders) | 5 | 2 | 7
Asthenia (General disorders) | 2 | 2 | 4
Mucosal inflammation (General disorders) | 1 | 1 | 2
Oedema peripheral (General disorders) | 0 | 1 | 1
Paronychia (Infections and infestations) | 3 | 1 | 4
Alveolar osteitis (Infections and infestations) | 2 | 0 | 2
Oral fungal infection (Infections and infestations) | 2 | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dry eye (Eye disorders) | 4 | 1 | 5
Weight decreased (Investigations) | 4 | 0 | 4
Dysgeusia (Nervous system disorders) | 2 | 0 | 2
Ageusia (Nervous system disorders) | 0 | 1 | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
Due to low rates of investigator and patient recruitment, it appeared that it would not be possible to recruit the target patient population in an acceptable timeframe and the study was prematurely stopped

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT02483416/Prot_SAP_000.pdf